CLINICAL TRIAL: NCT03669016
Title: Mindfulness for Students
Acronym: Mindfulstud
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Helsinki (Other)
Collaborators: University of Cambridge (Other); University of Jyvaskyla (Other); Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Saara Repo, Principal Investigator, Senior lecturer in University Pedagogy, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MIndfulness for Students
Record Dates: First submitted 2018-08-31; First posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Well-being; Functional Ability; Stress; Mindfulness
Keywords: well-being; functional ability; stress; mindfulness; undergaduate students

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Face-to-face group-based mindfulness (Experimental): 8 weeks training.
  Interventions: Behavioral: Face-to-face group-based mindfulness
- Internet-based mindfulness (Experimental): 8 weeks training.
  Interventions: Behavioral: Internet-based mindfulness
- Waiting-list control group (No Intervention): No training during the study.

INTERVENTIONS:
Behavioral: Face-to-face group-based mindfulness — An eight-week course, including 75-90 minutes once-a-week meeting. Participants are supposed to practice mindfulness skills in their spare time 10-30 minutes per day. An eight-week course, including 75-90 minutes once-a-week meeting. Participants are supposed to practice mindfulness skills in their spare time 10-30 minutes per day. This training is based on Jon Kabat-Zinn's course Mindfulness Based Stress Reduction and book Williams & Penman Mindfulness: a practical guide to finding peace in a frantic world and adapted for university students. In addition, a manual written in Cambridge University "Mindfulness Skills for Students" is utilized.
  Arms: Face-to-face group-based mindfulness
Behavioral: Internet-based mindfulness — An eight-week course, including 60 minutes starting and ending meeting. Participants are practicing mindfulness, doing other tasks (writing, reading, reflecting) on their own. This course is created in University of Jyväskylä, Finland. It is based on mindfulness and Acceptance and Commmitment Therapy.
  Arms: Internet-based mindfulness

SUMMARY:
The aim of the study is to find out, weather the students' wellbeing and functional ability can be enhanced by two different type of mindfulness interventions: 1) face-to-face group-based training, and 2) internet-based training based in mindfulness and acceptance and commitment therapy. Study results may be used to decide whether it is worth offering mindfulness training for medical faculty students, and what kind of training would be most suitable and effective in the medical education context.

DETAILED DESCRIPTION:
The hypotheses is that participating to the mindfulness intervention improves students well-being and decreases their level of stress. These are measured by self-evaluation questionnaires and with hair samples, before the intervention, immediately after intervention and four months after the intervention.

This is a randomized control trial. There are two different experiment groups and one waiting-list control group. The target group is all undergraduate students in the Faculty of Medicine, University of Helsinki. The participants are recruited with e-mail and informing students in different situations. The aimed amount of participants is 120-150 but the study will be conducted if 90 participants are recruited. The participants enroll to the study by signing consent format.

This is a follow-up research. The person register (name, university e-mail address, student number) are used to recruitment and to ensure the participants identity.

Time of data preservation is 10 years. The last student register data is going to be collected 2019. The data is preserved until age 2029.

The questionnaire with which the main data is been collected is Webropol questionnaire tool. The data is removed from the Webropol after three months of the end of the questionnaire answer time. The person responsible for the data removes the data from University's server after ten years.

Content of the register

1. Mindfulness for Students questionnaire data
2. Mindfulness for Students hair samples
3. Mindfulness for students -observation log
4. Mindfulness for students -interview data
5. Data collected in Student Compass -internet environment
6. Data of students' credits are collected from University's own credit register "Oodi", if participant has given a consent to that.

Students are being recruited in information meeting. They will be informed orally in that situation and given a written communication paper. The students who want to participate the course, will fill and sign a consent format. In format there is a research number code given to the student. The connection between the student identity and the research code number is known only by the persons that are responsible for the database.

ELIGIBILITY:
Inclusion Criteria:

- All undergraduate students of Faculty of Medicine, University of Helsinki who have started their studies in year 2009 or after that.

Exclusion Criteria:

* The participants that can not participate fully to the intervention (self-evaluated).
* Participants who have severe mental problems (like anxiety or depression) when the study starts,
* Participants who have hade a great loss or trauma in near past, or some other mental or physical health problem that could make participation difficult.

This is evaluated based on how the participants answers to the base line questionnaire the following measures:

1. answers to the CORE-OM questionnaire and
2. answers to the questions where participants evaluate themselves their anxiety, depression, mental health.
3. If participant tell they have some other mental disorder, they are not accepted to the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-08-22 (Actual); Primary Completion 2019-04-15 (Estimated); Study Completion 2019-04-15 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline CORE-OM measure at post-intervention and 4-month follow-up. | It is measured three weeks before the intervention starts, immediately after the 8-week intervention is finished, and 4-month after the intervention is finished.
  CORE-OM, Clinical Outcomes in Routine Evaluation Outcome Measure.

SECONDARY OUTCOMES:
Change from Baseline rate of stress at post-intervention and 4-month follow-up. | It is measured in the same day when the intervention starts, immediately after the 8-week intervention is finished, and 4-month after the intervention is finished.
  Cortisol as an indicator of stress which is measured from hair samples. Stadler & Kirschbaum 2012.
Change from Baseline rate of resilience in studies at post-intervention and 4-month follow-up. | It is measured three weeks before the intervention starts, immediately after the 8-week intervention is finished, and 4-month after the intervention is finished.
  Workplace Acceptance and Action Questionnaire (WAAQ) applied for students. Bond, Joda, and Guenole 2013; Asikainen, Hailikari, Mattson 2017.
Change from Baseline rate of social support in studies at post-intervention and 4-month follow-up. | It is measured three weeks before the intervention starts, immediately after the 8-week intervention is finished, and 4-month after the intervention is finished.
  Application of questionnaires of social support from Sarason et al. 1987 and Pyörälä et al. 2015.
Change from Baseline rate of study load in studies at post-intervention and 4-month follow-up. | It is measured three weeks before the intervention starts, immediately after the 8-week intervention is finished, and 4-month after the intervention is finished.
  Application of questionnaire of healthy work measure of Karasek & Theorell 1990.
Students' possibilities to influence to their own studies | It is measured three weeks before the interventions start.
  Application of measures of healthy work measure. Karasek & Theorell 1990.
Change from Baseline rate of functional ability in studies at post-intervention and 4-month follow-up. | It is measured three weeks before the intervention starts, immediately after the 8-week intervention is finished, and 4-month after the intervention is finished.
  Application of functional ability at work. Tuomi et al. 1998.
Change from Baseline rate of subjective experience of quality of life at post-intervention and 4-month follow-up. | It is measured three weeks before the intervention starts, immediately after the 8-week intervention is finished, and 4-month after the intervention is finished.
  Subjective experience of quality of life. One Likert-scale question adapted and modified from three different questionnaires. Koivumaa et al. 2000; Allardt 1973; Lundqvist & Mäkiopas 2016)
Change from Baseline rate of mental well-being Scale at post-intervention and 4-month follow-up. | It is measured three weeks before the intervention starts, immediately after the 8-week intervention is finished, and 4-month after the intervention is finished.
  The Warwick-Edinburgh Mental Well-being Scale
Change from Baseline rate of Personality at post-intervention and 4-month follow-up. | It is measured three weeks before the intervention starts, immediately after the 8-week intervention is finished, and 4-month after the intervention is finished.
  Parts of Big Five (Lang et al. 2011)
Change from Baseline rate of sense of coherence at post-intervention and 4-month follow-up. | It is measured three weeks before the intervention starts, immediately after the 8-week intervention is finished, and 4-month after the intervention is finished.
  Sence of coherence - SOC 3 (Antonovsky 1987; Schumann et al. 2003)
Change from Baseline rate of Resilience at post-intervention and 4-month follow-up. | It is measured three weeks before the intervention starts, immediately after the 8-week intervention is finished, and 4-month after the intervention is finished.
  Resilience scale (Wagnild & Young, 1993; Losoi et al 2013 modified)
Change from Baseline rate of experiences of own health at post-intervention and 4-month follow-up. | It is measured three weeks before the intervention starts, immediately after the 8-week intervention is finished, and 4-month after the intervention is finished.
  Questionnaire Kunttu et al. 2017
Change from Baseline rate of quality and length of sleep at post-intervention and 4-month follow-up. | It is measured three weeks before the intervention starts, immediately after the 8-week intervention is finished, and 4-month after the intervention is finished.
  Basic Nordic Sleep Questionnaire shortened (Partinen & Gislason 1995)
Change from Baseline rate of fatigue in day-time at post-intervention and 4-month follow-up. | It is measured three weeks before the intervention starts, immediately after the 8-week intervention is finished, and 4-month after the intervention is finished.
  Questionnaire from Health 2000/2001 Research in Finland
Change from Baseline amount of nightmares during previous month at post-intervention and 4-month follow-up. | IIt is measured three weeks before the intervention starts, immediately after the 8-week intervention is finished, and 4-month after the intervention is finished.
  Application of questionnaire Sandman et al 2015.
Participant's own evaluation of his/her mental health | Three weeks before the intervention starts
  Participant's own evaluation of the symptoms of mental health during previous month.
Change from Baseline approximate amount of exercise at post-intervention and 4-month follow-up. | It is measured three weeks before the intervention starts, immediately after the 8-week intervention is finished, and 4-month after the intervention is finished.
  Questionnaire from Health 2000/2001 Research in Finland
Change from Baseline regularity of eating habits at post-intervention and 4-month follow-up. | It is measured before intervention, post-intervention and 4-month follow-up.
  Participant's own evaluation of the regularity of eating habits.
Change from Baseline approximate amount of caffeine used daily. at post-intervention and 4-month follow-up. | IIt is measured three weeks before the intervention starts, immediately after the 8-week intervention is finished, and 4-month after the intervention is finished.
  Participant's own evaluation of the amount of daily caffeine use.
Change from Baseline approximate amount use of alcohol and cigarettes daily. | It is measured three weeks before the intervention starts, immediately after the 8-week intervention is finished, and 4-month after the intervention is finished.
  Participant's own evaluation of approximate amount use of alcohol and cigarettes daily.
Change from Baseline rate of Mindfulness skills at post-intervention and 4-month follow-up. | It is measured three weeks before the intervention starts, immediately after the 8-week intervention is finished, and 4-month after the intervention is finished.
  Freiburg Mindfulness Index (FMI) Walach, H., Buchheld, N., Buttenmüller, V., Kleinknecht, N., & Schmidt, S. 2006; Lehto, Uusitalo-Malmivaara & Repo 2015.
Change from Baseline rate of stress and recovery of it at post-intervention and 4-month follow-up. | IIt is measured three weeks before the intervention starts, immediately after the 8-week intervention is finished, and 4-month after the intervention is finished.
  Application of measures of healthy work measure of Lundqvist & Mäkiopas 2016 and Elo et al. 1992.
Previous experience in practicing of mindfulness and/or meditation | It is measured three weeks before the intervention starts.
  Participant's own evaluation of the amount of previous experience in practicing mindfulness and/or meditation
Amount and quality of independent mindfulness practice | Immediately after the 8-week intervention is finished.
  Participant's self-evaluation of amount and quality of independent mindfulness practice
Change from post-intervention amount and quality of independent mindfulness practice at 4-month follow-up. | Immediately after the 8-week intervention is finished, and 4-month after the intervention is finished.
  Participant's self-evaluation of amount and quality of independent mindfulness practice.

CONTACTS AND LOCATIONS:
Overall Officials: Saara Repo, PhD, Principal Investigator — University of Helsinki
Locations (1):
- University of Helsinki, Helsinki, University of Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Miller R, Wankerl M, Stalder T, Kirschbaum C, Alexander N. The serotonin transporter gene-linked polymorphic region (5-HTTLPR) and cortisol stress reactivity: a meta-analysis. Mol Psychiatry. 2013 Sep;18(9):1018-24. doi: 10.1038/mp.2012.124. Epub 2012 Sep 4. PMID 22945032
- [Background] Daya Z, Hearn JH. Mindfulness interventions in medical education: A systematic review of their impact on medical student stress, depression, fatigue and burnout. Med Teach. 2018 Feb;40(2):146-153. doi: 10.1080/0142159X.2017.1394999. Epub 2017 Nov 7. PMID 29113526
- [Result] Galante J, Dufour G, Vainre M, Wagner AP, Stochl J, Benton A, Lathia N, Howarth E, Jones PB. A mindfulness-based intervention to increase resilience to stress in university students (the Mindful Student Study): a pragmatic randomised controlled trial. Lancet Public Health. 2018 Feb;3(2):e72-e81. doi: 10.1016/S2468-2667(17)30231-1. Epub 2017 Dec 19. PMID 29422189
- [Derived] Kunzler AM, Helmreich I, Konig J, Chmitorz A, Wessa M, Binder H, Lieb K. Psychological interventions to foster resilience in healthcare students. Cochrane Database Syst Rev. 2020 Jul 20;7(7):CD013684. doi: 10.1002/14651858.CD013684. PMID 32691879